CLINICAL TRIAL: NCT00365365
Title: A Phase IIb, Randomized, Multicenter, Noncomparative Pilot Study of the Safety & Efficacy of Three Docetaxel-Based Chemotherapy Regimens Plus Bevacizumab ± Trastuzumab for the Adjuvant Treatment of Patients With Node-Positive & High-Risk Node-Negative Breast Cancer
Brief Title: Safety & Efficacy of Three Docetaxel-Based Chemotherapy Regimens Plus Bevacizumab With or Without Trastuzumab for Adjuvant Treatment of Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_00714
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Bevacizumab; Docetaxel; Carboplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stratum 1 (AC->T + bevacizumab) (Experimental): HER2-negative participants administered
  * doxorubicin and cyclophosphamide (AC) + bevacizumab for 4 cycles followed by
  * docetaxel (T) + bevacizumab for 4 cycles followed by
  * bevacizumab maintenance therapy for total of 52 weeks from date of first dose regardless of number of doses received or missed
  Interventions: Drug: Doxorubicin and cyclophosphamide (AC) + bevacizumab; Drug: Docetaxel (T) + bevacizumab; Drug: Bevacizumab maintenance therapy
- Stratum 2 (TAC + bevacizumab) (Experimental): HER2-negative participants administered
  * docetaxel, doxorubicin, cyclophosphamide (TAC) + bevacizumab for 6 cycles followed by
  * bevacizumab maintenance therapy for total of 52 weeks from date of first dose regardless of number of doses received or missed
  Interventions: Drug: Docetaxel, doxorubicin, cyclophosphamide (TAC) + bevacizumab; Drug: Bevacizumab maintenance therapy
- Stratum 3 (TCH + bevacizumab) (Experimental): All HER2-positive participants administered
  * docetaxel, carboplatin, trastuzumab (TCH) + bevacizumab for 6 cycles followed by
  * bevacizumab and trastuzumab maintenance therapy for total of 52 weeks from date of first dose regardless of number of doses received or missed
  Interventions: Drug: Docetaxel, carboplatin, trastuzumab (TCH) + bevacizumab; Drug: Bevacizumab and trastuzumab maintenance therapy

INTERVENTIONS:
Drug: Doxorubicin and cyclophosphamide (AC) + bevacizumab — For every 3-week cycle
  * bevacizumab 15 mg/kg infused intravenously (IV) on Day 1 followed by
  * doxorubicin 60 mg/m^2 IV push or infusion followed by cyclophosphamide 600 mg/m^2 IV push or infusion
  * Prophylactic G-CSF was administered within 24 hours following each cycle of chemotherapy but no greater than 72 hours after chemotherapy
  Other Names: Avastin® (bevacizumab); Adriamycin® (doxorubicin)
  Arms: Stratum 1 (AC->T + bevacizumab)
Drug: Docetaxel (T) + bevacizumab — For every 3-week cycle
  * bevacizumab 15 mg/kg infused intravenously (IV) on Day 1 followed by
  * docetaxel 100 mg/m^2 IV
  * Prophylactic G-CSF was administered within 24 hours following each cycle of chemotherapy but no greater than 72 hours after chemotherapy
  Note: The starting dose of docetaxel was reduced to 75 mg/m^2 if toxicity occurred that met the criteria for doxorubicin dose reduction
  Other Names: Taxotere® (docetaxel); Avastin® (bevacizumab)
  Arms: Stratum 1 (AC->T + bevacizumab)
Drug: Docetaxel, doxorubicin, cyclophosphamide (TAC) + bevacizumab — For every 3-week cycle
  * bevacizumab 15 mg/kg infused intravenously (IV) on Day 1 followed by
  * doxorubicin 50 mg/m^2 IV push or infusion followed by cyclophosphamide 500 mg/m^2 IV push or infusion followed by docetaxel 75 mg/m^2
  * Prophylactic G-CSF was administered within 24 hours following each cycle of chemotherapy but no greater than 72 hours after chemotherapy
  Other Names: Taxotere® (docetaxel); Avastin® (bevacizumab)
  Arms: Stratum 2 (TAC + bevacizumab)
Drug: Docetaxel, carboplatin, trastuzumab (TCH) + bevacizumab — For every 3-week cycle
  * bevacizumab 15 mg/kg infused intravenously (IV) on Day 1 followed by
  * docetaxel in 75 mg/m^2 IV followed by carboplatin AUC 6 mg/mL/min IV followed by
  * trastuzumab 6 mg/kg by IV infusion (For the first cycle 1 only a loading dose of trastuzumab 8 mg/kg IV was infused on Day 2)
  * Prophylactic G-CSF was administered within 24 hours following each cycle of chemotherapy but no greater than 72 hours after chemotherapy
  Other Names: Taxotere® (docetaxel); Herceptin® (trastuzumab); Avastin® (bevacizumab)
  Arms: Stratum 3 (TCH + bevacizumab)
Drug: Bevacizumab and trastuzumab maintenance therapy — * bevacizumab 15 mg/kg was infused IV followed by
  * trastuzumab 6 mg/kg IV
  Treatment was every 3 weeks for 52 weeks from the date of the first administration regardless of the number of doses received or missed.
  Other Names: Avastin® (bevacizumab); Herceptin® (trastuzumab)
  Arms: Stratum 3 (TCH + bevacizumab)
Drug: Bevacizumab maintenance therapy — - bevacizumab 15 mg/kg was infused IV
  Treatment was every 3 weeks for 52 weeks from the date of the first administration regardless of the number of doses received or missed.
  Other Names: Avastin® (bevacizumab)
  Arms: Stratum 1 (AC->T + bevacizumab); Stratum 2 (TAC + bevacizumab)

SUMMARY:
This is a phase IIb, randomized, parallel-group, noncomparative, multicenter, pilot study designed to evaluate the safety and efficacy of bevacizumab with or without (+/-) trastuzumab administered with three different docetaxel-based combination regimens for the adjuvant treatment of participants with node positive or high-risk node negative breast cancer.

DETAILED DESCRIPTION:
In this study, participants were stratified according to HER2 status at the time of enrollment. HER2-negative participants were randomized in a 1:1 ratio to either stratum 1 (AC->T sequential + bevacizumab) or stratum 2 (TAC + bevacizumab). All HER2-positive participants were assigned to stratum 3 (TCH + bevacizumab).

The study included a treatment period of 1 year, followed by a 2 year posttreatment survival follow-up period.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow participants and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Inclusion Criteria:

* Women >/= 18 years of age.
* Histologically proven breast cancer with an interval between definitive breast surgery that includes axillary lymph node (LN) dissection or axillary nodal evaluation and study registration of < 60 days. (Note: Cycle 1 of chemotherapy treatment may NOT be infused until > 28 days after the date of definitive breast surgery and the participant must be recovered from any clinically significant toxicity thereof.)
* Definitive surgical treatment must be either mastectomy, or breast conserving surgery with axillary lymph node dissection (axillary lymph node evaluation can be either full axillary node dissection or sentinel LN evaluation followed by dissection if sentinel LN is positive) for operable breast cancer (pT1-4 [including inflammatory], pNO-3, and MO). Margins of resected specimen from definitive surgery must be histologically free of invasive adenocarcinoma and ductal carcinoma in-situ (DCIS). Lobular carcinoma in-situ does not count as a positive margin.
* Subjects must be either lymph node-positive (pN1-3) or lymph node-negative (pN0) with high-risk features as determined by Investigator.
* High-risk, lymph node-negative participants, (pN0) will be defined as subjects having invasive adenocarcinoma with either a negative sentinel node biopsy (pN0[sn]) OR negative lymph node dissection (pN0) disease AND tumor size > 2 cm or tumor size >/= 1 cm with at least one of the following factors:

  * negative estrogen receptor (ER) and negative progesterone receptor (PR) status
  * histologic and/or nuclear Grade 2-3; or
  * age < 35 years
* HER2/neu positive or negative tumors are eligible. HER2 positivity must be documented by fluorescence in situ hybridization (FISH).
* Estrogen and progesterone receptor status must be performed on the primary tumor prior to study entry. Results must be pending or known at the time of study entry.
* Normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF) or shortening fraction (multiple-gated acquisition [MUGA] scan or echocardiography respectively). The result must be greater than the lower limit of normal (LLN) for the institution.
* Hematology evaluation within 2 weeks prior to study entry:

  * Absolute neutrophil count (ANC) >/= 1,500/μL
  * Platelets >/= 100,000/μL
  * Hemoglobin >/= 9 g/dL
* Hepatic function evaluation within 2 weeks prior to study entry:

  * Total bilirubin </= ULN for the institution
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be in the acceptable range.
* Complete staging work-up as follows: All subjects must have an appropriate radiographic evaluation, e.g., computed tomography (CT), positron emission tomography (PET)/CT, and/or (magnetic resonance imaging) MRI of the brain, chest, abdomen and pelvis, and imaging of bone by either a bone scan or PET scan. In cases of positive bone imaging, a bone X-ray or MRI evaluation is mandatory to rule out the possibility of metastatic bone scan disease. Other tests may be performed as clinically indicated. It is recommended that all baseline staging should be completed within 35 days prior to study entry.

Exclusion Criteria:

* Prior systemic anticancer therapy for breast cancer (immunotherapy, hormonotherapy, chemotherapy).
* Prior anthracycline therapy, taxoids or platinum salts for any malignancy.
* Prior radiation therapy for breast cancer or any radiotherapy to the chest wall for any other malignancy.
* Bilateral invasive breast cancer.
* Pregnant or lactating subjects
* Cardiac disease or risk for same as judged by Investigator
* Other serious illness or medical conditions such as (partial list- review with Investigator) history of significant neurologic or psychiatric disorders that would prohibit the understanding and giving of informed consent, active uncontrolled infection, active peptic ulcer, unstable diabetes mellitus or subjects with symptomatic, intrinsic lung disease resulting in dyspnea at rest
* Current therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (SERMs), either for osteoporosis or prevention of breast cancer. Subjects must have discontinued these agents prior to study entry.
* Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment must be stopped prior to study entry.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational non-marketed drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.
* Male subjects, as no clinical efficacy or safety data are available from phase I-II studies.
* Chemotherapy and/or bevacizumab may not be given until > 7 days following a minor surgical procedure. Chemotherapy may be given without bevacizumab in circumstances in which the participant has recovered sufficiently to receive chemotherapy but has not yet reached a 28 day time point at which bevacizumab could be administered.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2006-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Erickson, MSN, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 239 participants were screened in this study. 214 were considered eligible for enrollment and 25 were screen failures. Of the 214 eligible participants, 155 were HER2-negative and 59 were HER2-positive.
Groups:
- Stratum 3 (TCH + Bevacizumab).): All HER2-positive participants administered
  * docetaxel, carboplatin, trastuzumab (TCH) + bevacizumab for 6 cycles followed by
  * bevacizumab and trastuzumab maintenance therapy for total of 52 weeks from date of first dose regardless of number of doses received or missed
Period: Overall Study
Arm/Group | Stratum 1 (AC->T + Bevacizumab) | Stratum 2 (TAC + Bevacizumab) | Stratum 3 (TCH + Bevacizumab).)
Started | 78 | 77 | 59
TREATED (SAFETY POPULATION) | 78 | 75 | 59
COMPLETED TREATMENT | 38 | 36 | 45
Completed | 44 | 41 | 44
Not Completed | 34 | 36 | 15
Not completed — Randomized but not treated | 0 | 2 | 0
Not completed — Poor compliance to protocol | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Death | 1 | 3 | 0
Not completed — Subject's request | 11 | 13 | 1
Not completed — Disease progression/relapse | 9 | 6 | 7
Not completed — Adverse Event | 6 | 6 | 3
Not completed — Moved | 2 | 0 | 0
Not completed — New cancer | 1 | 0 | 0
Not completed — Withdrew consent | 1 | 1 | 0
Not completed — Second malignancy | 0 | 1 | 0
Not completed — Patient/physician decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 (AC->T + Bevacizumab) | Stratum 2 (TAC + Bevacizumab) | Stratum 3 (TCH + Bevacizumab).) | Total
Number analyzed (Participants) | 78 | 75 | 59 | 212
Age Continuous [Mean (Standard Deviation); unit: years] | 53.0 (10.45) | 55.1 (9.89) | 50.8 (9.61) | 53.1 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 59 | 212
  Male | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group Score (ECOG) [Number; unit: participants] — The ECOG score assesses how the disease affects a participant's daily living abilities. It ranges from 0-5, with 0 being the best and 5 being the worst outcome. "0" reflects a fully active participant, able to carry on all pre-disease performance without restriction. "1" reflects a participant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  participants
    ECOG Score = 0 | 73 | 67 | 55 | 195
    ECOG Score = 1 | 5 | 8 | 4 | 17
Electrocardiogram (ECG) [Number; unit: participants] — Electrocardiogram (ECG) findings were reported.
  participants
    Normal | 45 | 53 | 36 | 134
    Abnormal | 22 | 19 | 19 | 60
    Not done/missing | 11 | 3 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Safety - Number of Participants With Grade 3-4 Clinical Congestive Heart Failure (CHF)
Description: Participants were evaluated for clinical CHF every 3 weeks during chemotherapy, every 3 months while on maintenance therapy, and every 3 months during the 2-year follow-up period. Left ventricular ejection fraction (LVEF) of CHF was assessed by multi-gated acquisition (MUGA) or echocardiogram (ECHO) performed midway through completion of chemotherapy according to a treatment-specific schedule, every 12 weeks during maintenance therapy, and at 6 and 24 months after completion of maintenance therapy.
  Grade 3-4 CHF were identified through a clinical review of all study collected investigator verbatim and the Medical Dictionary for Regulatory Activities (MedDRA). The preferred terms (PT) cardiac failure congestive, cardiomyopathy, and ejection fraction decreased were associated with CHF.
Time Frame: from the first dose of study medication up to the end of follow-up (up to 3 yrs)
Population: Safety population - participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Stratum 1 (AC->T + Bevacizumab) | Stratum 2 (TAC + Bevacizumab) | Stratum 3 (TCH + Bevacizumab).)
Number analyzed (Participants) | 78 | 75 | 59
participants | 1 [0.0 to 6.9] | 3 [0.8 to 11.2] | 1 [0.0 to 0.1]

2. Secondary Outcome: Safety - Number of Participants With Adverse Events (AE)
Description: An adverse event was any untoward medical occurrence in a participant of the clinical investigation, regardless of the relationship to study treatment.
  A serious adverse event (SAE) was an AE that at any dose (including overdose) resulted in death, was life-threatening, required inpatient hospitalization or prolonged existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly/birth defect, and/or was medically important.
  Treatment-emergent adverse events (TEAE) were defined as AEs that developed or worsened in severity during the on-treatment period.
Time Frame: from the administration of the first dose of study medication up to 30 days after the last dose of study medication; events ongoing at the time of discontinuation were monitored in the follow-up period until resolution.
Population: Safety population - participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Stratum 1 (AC->T + Bevacizumab) | Stratum 2 (TAC + Bevacizumab) | Stratum 3 (TCH + Bevacizumab).)
Number analyzed (Participants) | 78 | 75 | 59
participants
  with TEAE | 78 | 75 | 59
  with serious TEAE | 23 | 24 | 12
  with any TEAE leading to death | 0 | 2 | 0
  with any TEAE leading to treatment discontinuation | 21 | 24 | 16
  with any Grade 3-4 Serious TEAE | 23 | 24 | 9

3. Secondary Outcome: Disease-free Survival (DFS) Rate
Description: DFS was defined as the time from the administration of the first-dose of study medication until recurrence of tumor or death from any cause in the absence of previous documentation of tumor recurrence. DFS rate was the probability of being disease free and alive at a particular time. DFS rates were estimated using Kaplan-Meier Method, and 95% confidence intervals were computed using the method of Kalbfleisch and Prentice.
  For participants who did have objective recurrence of tumor and who were still on study at the time of an analysis, or who were given antitumor treatment other than the study treatment, or who were removed from study follow-up prior to documentation of the tumor recurrence, DFS was censored at the last date the participant was known to be disease-free.
Time Frame: from the administration of the first-dose of study medication up to 12 months, 18 months and 24 months
Population: Intent-to-treat population - All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: Number of DFS events
Arm/Group | Stratum 1 (AC->T + Bevacizumab) | Stratum 2 (TAC + Bevacizumab) | Stratum 3 (TCH + Bevacizumab).)
Number analyzed (Participants) | 78 | 77 | 59
Number analyzed (Number of DFS events) | 10 | 9 | 7
percentage of participants
  DFS rate at 12 months | 93.6 [83.8 to 97.5] | 95.9 [87.8 to 98.7] | 98.2 [87.8 to 99.7]
  DFS rate at 24 months | 87.1 [75.9 to 93.4] | 94.1 [84.8 to 97.8] | 96.3 [86.0 to 99.1]
  DFS rate at 36 months | 85.5 [74.0 to 92.2] | 90.4 [79.6 to 95.6] | 90.4 [78.5 to 95.9]

ADVERSE EVENTS:
Groups:
- AC->T + Bevacizumab: HER2-negative participants administered
  * doxorubicin and cyclophosphamide (AC) + bevacizumab for 4 cycles followed by
  * docetaxel (T) + bevacizumab for 4 cycles followed by
  * bevacizumab maintenance therapy for total of 52 weeks from date of first dose regardless of number of doses received or missed
- TAC + Bevacizumab: HER2-negative participants administered
  * docetaxel, doxorubicin, cyclophosphamide (TAC) + bevacizumab for 6 cycles followed by
  * bevacizumab maintenance therapy for total of 52 weeks from date of first dose regardless of number of doses received or missed
- TCH + Bevacizumab: All HER2-positive participants administered
  * docetaxel, carboplatin, trastuzumab (TCH) + bevacizumab for 6 cycles followed by
  * bevacizumab and trastuzumab maintenance therapy for total of 52 weeks from date of first dose regardless of number of doses received or missed
Arm/Group | AC->T + Bevacizumab | TAC + Bevacizumab | TCH + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 23/78 | 24/75 | 12/59
Other Adverse Events (participants affected / at risk) | 78/78 | 75/75 | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AC->T + Bevacizumab (N=78) | TAC + Bevacizumab (N=75) | TCH + Bevacizumab (N=59)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Incision site abscess (Infections and infestations) | 0 | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AC->T + Bevacizumab (N=78) | TAC + Bevacizumab (N=75) | TCH + Bevacizumab (N=59)
Anaemia (Blood and lymphatic system disorders) | 45 | 42 | 32
Neutropenia (Blood and lymphatic system disorders) | 41 | 41 | 8
Leukopenia (Blood and lymphatic system disorders) | 33 | 35 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 37 | 29
Lymphopenia (Blood and lymphatic system disorders) | 8 | 8 | 3
Leukocytosis (Blood and lymphatic system disorders) | 4 | 6 | 1
Granulocytosis (Blood and lymphatic system disorders) | 3 | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 8 | 0
Tachycardia (Cardiac disorders) | 4 | 12 | 3
Ear pain (Ear and labyrinth disorders) | 6 | 3 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 3
Lacrimation increased (Eye disorders) | 29 | 8 | 17
Vision blurred (Eye disorders) | 6 | 1 | 3
Visual impairment (Eye disorders) | 4 | 2 | 1
Blepharospasm (Eye disorders) | 0 | 4 | 3
Nausea (Gastrointestinal disorders) | 64 | 60 | 51
Constipation (Gastrointestinal disorders) | 40 | 29 | 30
Diarrhoea (Gastrointestinal disorders) | 39 | 48 | 38
Vomiting (Gastrointestinal disorders) | 32 | 31 | 23
Dyspepsia (Gastrointestinal disorders) | 20 | 16 | 12
Stomatitis (Gastrointestinal disorders) | 19 | 17 | 7
Dysphagia (Gastrointestinal disorders) | 12 | 9 | 4
Dry mouth (Gastrointestinal disorders) | 11 | 5 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 10 | 4
Abdominal pain (Gastrointestinal disorders) | 8 | 18 | 12
Oesophagitis (Gastrointestinal disorders) | 8 | 0 | 1
Oral pain (Gastrointestinal disorders) | 8 | 8 | 9
Gingival bleeding (Gastrointestinal disorders) | 6 | 7 | 3
Abdominal discomfort (Gastrointestinal disorders) | 5 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4 | 5
Haemorrhoids (Gastrointestinal disorders) | 5 | 2 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 3 | 7
Abdominal distension (Gastrointestinal disorders) | 4 | 4 | 4
Haematochezia (Gastrointestinal disorders) | 3 | 2 | 5
Mouth ulceration (Gastrointestinal disorders) | 3 | 3 | 6
Fatigue (General disorders) | 71 | 61 | 51
Mucosal inflammation (General disorders) | 37 | 16 | 15
Pyrexia (General disorders) | 21 | 24 | 15
Oedema peripheral (General disorders) | 16 | 11 | 7
Asthenia (General disorders) | 15 | 20 | 11
Pain (General disorders) | 13 | 5 | 6
Chills (General disorders) | 10 | 5 | 7
Oedema (General disorders) | 6 | 4 | 6
Catheter site pain (General disorders) | 4 | 5 | 4
Influenza like illness (General disorders) | 4 | 2 | 3
Tenderness (General disorders) | 3 | 1 | 3
Chest discomfort (General disorders) | 2 | 2 | 7
Seasonal allergy (Immune system disorders) | 4 | 2 | 3
Candidiasis (Infections and infestations) | 12 | 4 | 1
Sinusitis (Infections and infestations) | 8 | 9 | 10
Nasopharyngitis (Infections and infestations) | 7 | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 7
Urinary tract infection (Infections and infestations) | 7 | 14 | 10
Oral candidiasis (Infections and infestations) | 6 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 2 | 0
Catheter site infection (Infections and infestations) | 2 | 0 | 3
Pharyngitis (Infections and infestations) | 2 | 2 | 3
Bronchitis (Infections and infestations) | 1 | 5 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 12 | 9 | 9
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 4
Weight decreased (Investigations) | 9 | 10 | 5
Aspartate aminotransferase increased (Investigations) | 8 | 3 | 7
Alanine aminotransferase increased (Investigations) | 7 | 3 | 7
Ejection fraction decreased (Investigations) | 5 | 7 | 7
Blood pressure increased (Investigations) | 4 | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 6
Haemoglobin decreased (Investigations) | 3 | 1 | 5
Platelet count decreased (Investigations) | 2 | 3 | 4
Blood glucose increased (Investigations) | 1 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 39 | 25 | 22
Dehydration (Metabolism and nutrition disorders) | 20 | 17 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 9 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 51 | 37 | 32
Myalgia (Musculoskeletal and connective tissue disorders) | 38 | 23 | 21
Bone pain (Musculoskeletal and connective tissue disorders) | 22 | 23 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 15 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 16 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 7 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 4 | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Headache (Nervous system disorders) | 37 | 26 | 24
Neuropathy peripheral (Nervous system disorders) | 20 | 8 | 12
Dysgeusia (Nervous system disorders) | 18 | 19 | 18
Dizziness (Nervous system disorders) | 13 | 12 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 7 | 5
Hypoaesthesia (Nervous system disorders) | 7 | 4 | 5
Sinus headache (Nervous system disorders) | 7 | 2 | 1
Paraesthesia (Nervous system disorders) | 5 | 6 | 6
Migraine (Nervous system disorders) | 3 | 2 | 3
Insomnia (Psychiatric disorders) | 30 | 30 | 16
Anxiety (Psychiatric disorders) | 16 | 13 | 9
Depression (Psychiatric disorders) | 10 | 10 | 11
Proteinuria (Renal and urinary disorders) | 14 | 12 | 11
Dysuria (Renal and urinary disorders) | 6 | 3 | 2
Haematuria (Renal and urinary disorders) | 2 | 6 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 1 | 3
Breast pain (Reproductive system and breast disorders) | 2 | 6 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 36 | 32 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32 | 21 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 15 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 14 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 58 | 48 | 50
Nail disorder (Skin and subcutaneous tissue disorders) | 23 | 3 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 16 | 10 | 20
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6 | 5 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 9 | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Sinus operation (Surgical and medical procedures) | 9 | 6 | 5
Hot flush (Vascular disorders) | 25 | 18 | 12
Hypertension (Vascular disorders) | 23 | 21 | 16
Lymphoedema (Vascular disorders) | 12 | 8 | 5
Flushing (Vascular disorders) | 2 | 5 | 5

LIMITATIONS AND CAVEATS:
The study was originally designed to last for 6-10 years. Based on a protocol amendment, the study was shortened to about 3 years, and the endpoint Overall Survival (OS) was deleted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days for abstracts) in advance of any submission for publication. The Sponsor may request for the publication to be delayed for upto 90 days to preserve its proprietary rights.